CLINICAL TRIAL: NCT05925855
Title: Effect of Phonophoresis on Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Reem Dawood, Assistant professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phonophoresis
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2023-07

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — ketoprofen topical gel; Escin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- study Fastum (Experimental): participant in this group will receive US with fastum gel
  Interventions: Other: US with fastum
- study Reparil (Experimental): participant in this group will receive US with reparil gel
  Interventions: Other: US with reparil
- Control plain gel (Active Comparator): participant in this group will receive US with gel
  Interventions: Other: US with plain gel

INTERVENTIONS:
Other: US with fastum — apply fastum on trigger point with US
  Arms: study Fastum
Other: US with reparil — apply reparil on trigger point with US
  Arms: study Reparil
Other: US with plain gel — apply gel on trigger point with US
  Arms: Control plain gel

SUMMARY:
purpose of this study was to investigate the effects of phonophoresis with fastum gel versus reparil gel on pain intensity, pain threshold, and cervical ROM of participant with trigger point of upper trapezius.

DETAILED DESCRIPTION:
participants will be divided into 3 groups, 2 study groups and 1 control group.

ELIGIBILITY:
Inclusion Criteria:

* upper trapezius trigger point

Exclusion Criteria:

* cervical disc

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | Two weeks
  change of pain intensity by using VAS from 0 to 10
pain threshold | two weeks
  change of pain threshold by using PPA
ROM | two weeks
  change of ROM by using CROM

CONTACTS AND LOCATIONS:
Overall Officials: Osama R Abdelraouf, PhD, Study Director — Batterjee Medical College
Locations (1):
- Batterjee Medical College, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
all data are secured with principle investigator.